## **Cover Page**

Title: Primary Cecal Pathologies Presenting as Acute Abdomen and Critical Appraisal of Their

Current Management Strategies in Emergency Settings

NCT Identifier Number: Not assigned

**Document Date:** 01/01/2016

## **Informed Consent for Participation in Study**

| I agree to get my patient to be part of this study at Jawaharlal Nehru Medical College, Aligarh |
|---|
| Muslim University, Aligarh. The effect and nature of operation and anaesthesia and associated |
| risks have been explained to me. |
| Signature of Patient's Attendant: |
| Date of Consent: |
| Consent verified by (Name, Designation and Signature): |